CLINICAL TRIAL: NCT06022432
Title: Overcoming Treatment Barriers: The Role of Expectations in the Behavioral Intention of Treatment Seeking for Social Anxiety
Brief Title: Overcoming Treatment Barriers
Acronym: OBSTACLE-S
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philipps University Marburg (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-76k
Record Dates: First submitted 2023-06-22; First posted 2023-09-01 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Health Care Utilization; Health Care Seeking Behavior
MeSH Terms: conditions — Patient Acceptance of Health Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Reducing Negative Expectations (Experimental): This group will watch a video of a patient-therapist interaction. The testimonial of the patient is framed to reduce negative expectations about therapeutic treatment.
  Interventions: Other: Video of a patients testimonial
- Maximizing Positive Expectations (Experimental): This group will watch a video of a patient-therapist interaction. The testimonial of the patient is framed to maximize positive expectations about therapeutic treatment.
  Interventions: Other: Video of a patients testimonial
- Control Group (Other): This group will explicate their current treatment expectations in a writing task.
  Interventions: Other: Writing Task

INTERVENTIONS:
Other: Video of a patients testimonial — The intervention is a prerecorded video of a re-enacted patient-therapist interaction whereby the patient gives a testimonial about the treatment process while either reducing negative expectations or maximizing positive expectations about therapy, respectively.
  Other Names: Free-Writing Task
  Arms: Maximizing Positive Expectations; Reducing Negative Expectations
Other: Writing Task — Participants write freely about their current treatment expectations / apprehensions to seek treatment
  Arms: Control Group

SUMMARY:
This study aims to assess whether negative or rather the lack of positive treatment expectations could be positively influenced by online short interventions and increase intention so seek treatment and actual help-seeking behavior when compared to a no-treatment control group. Further, the study investigators like to explore if specifically focusing on intensifying positive treatment expectations vs. a reduction of expectations about negative treatment effects will influence the pattern of results differently.

DETAILED DESCRIPTION:
The investigators expect that participants receiving an intervention e.g., amplifying positive (performance) expectancies vs. reducing negative (performance) expectancies of psychotherapeutic treatment, will show an increase in intentions to seek treatment and are more likely to report actual treatment-seeking behavior after the intervention when compared with participants who will describe their treatment expectations via a writing task.

Further, the investigators want to explore if the expectancy-modulating interventions will differently affect the intention to seek treatment within socially anxious individuals.

If participants agree, the investigators plan to assess changes in expectations, attitudes as well as actual treatment seeking behavior at a Follow-Up assessment one week later (data from Follow-Up will be analyzed exploratively and is not part of the main hypotheses).

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years old
* fluent in German (C Level)
* access to a computer device with internet access

Exclusion Criteria:

* non correctable hearing or visual impairment
* current in psychotherapeutic treatment or on a waiting list
* no neurological impairment or psychotic disorders

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2023-03-17 (Actual); Primary Completion 2024-02-15 (Actual); Study Completion 2024-06-13 (Actual)

PRIMARY OUTCOMES:
Change in Treatment Expectations (Treatment Expectation Questionnaire, "TEX-Q") | At baseline (pre-measurement), immediately after intervention (post-measurement, approximately 20 minutes after beginning of study procedure) and at Follow-Up investigation (one week after post measurement)
  Explicit treatment expectations measured by 15 items on a 11point Likert-scale
Changes in intention to seek treatment | At baseline (pre-measurement), immediately after intervention (post-measurement, approximately 20 minutes after beginning of study procedure) and at Follow-Up investigation (one week after post measurement)
  Estimated Probability to seek treatment on a self-generated rating scale from 0 (not likely at all) to 100 (very much likely)

SECONDARY OUTCOMES:
Intention to seek treatment (Behavioral Outcome 1) | After intervention (post measurement, approximately 30 minutes after beginning of study procedure)
  Participants respond with "yes" or "no" to indicate their interest to receive more concrete information about social anxiety and its treatment possibilities. If the answer was answered with "yes", participants are asked to give their e-mail address to receive information which is used to assess intention to seek treatment in form of a behavioral outcome.

OTHER OUTCOMES:
Treatment-seeking behavior (Behavioral Outcome 2) | At Follow-Up investigation (one week after post measurement)
  If participants agree to participate at our Follow Up, a second behavioral outcome will be assessed. Participants will be asked if they meanwhile have researched more concrete information about social anxiety online, connected with internet platforms or self-support groups, applied for online therapy programs/sessions, contacted or sought professional help for outpatient or psychiatric clinics. All categories have to be answered by a dichotomous scale ("yes" or "no").

CONTACTS AND LOCATIONS:
Locations (1):
- Philipps-Universität Marburg, Marburg, Germany

IPD SHARING:
Plan to Share IPD: No